CLINICAL TRIAL: NCT06847009
Title: Effect of Acupressure on Sleep Quality in Hemodialysis Patients: a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Didem Lafci (Other)
Responsible Party: Sponsor-Investigator, Didem Lafci, Asst. Prof. Dr., Mersin University
Organization: Mersin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mersin Ü.
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Hemodialysis Treatment; Acupressure; Sleep
Keywords: Hemodialysis Treatment; Patient; Nurse; Acupressure Application; Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: This study is single-blind, meaning that participants are unaware of whether they are in the intervention or control group, while care providers and investigators have access to this information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupressure Application Group (Experimental): This group consists of patients who have received acupressure. Acupressure will be applied to hemodialysis patients within the first two hours of HD and three times a week for four weeks. This intervention is carried out to evaluate sleep quality.
  Interventions: Other: Acupressure application
- Control Group (No Intervention): Routine nursing care will be applied to this group without acupressure. Additionally, measurements will be made regarding sleep quality.

INTERVENTIONS:
Other: Acupressure application — Acupressure will be applied to hemodialysis patients within the first two hours of HD and three times a week for four weeks. This intervention aims to evaluate its effects on sleep quality.
  Arms: Acupressure Application Group

SUMMARY:
This study aimed to evaluate the effects of acupressure applied to patients receiving hemodialysis treatment on sleep quality.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a common chronic disease worldwide and in our country, significantly affecting individuals' quality of life in physical, social, and psychological aspects. CKD is defined as a chronic and progressive deterioration of the kidney's fluid-solute balance and metabolic-endocrine functions due to the persistent decline in glomerular filtration rate (GFR) (Ammirati et al., 2020; Kalantar-Zadeh et al., 2021). Patients with a GFR below 5-10 ml/min require Renal Replacement Therapy (RRT). RRT is defined as a treatment method that replaces the kidney's normal blood filtration function when the kidneys can no longer perform this role. In the early stages of CKD, RRT becomes necessary when the disease cannot be controlled with diet and medication. Renal replacement therapies include hemodialysis, peritoneal dialysis, and renal transplantation (Tolasa et al., 2017; Eminsoy, 2018).

In our country, hemodialysis is the most preferred renal replacement therapy method for CKD treatment. The goal of hemodialysis is to improve patients' quality of life while reducing mortality and morbidity rates. Hemodialysis is a process in which blood is drawn from the patient through a suitable vascular access due to kidney failure, passed through a dialyzer (filter) with a semi-permeable membrane using a dialysis machine, and returned to the patient after removing waste substances such as urea, creatinine, and phosphorus from the blood (Webster et al., 2017; Yılmaz et al., 2020). Although hemodialysis helps control CKD-related complications, the treatment's dependency on a machine and its associated side effects-such as insomnia, fatigue, and restless legs syndrome-can negatively affect patients' quality of life (Merlino et al., 2006; Al-Jahemodiyalizali et al., 2010; Eminsoy, 2018; Hintistan et al., 2018; Tuna et al., 2018; Turgay et al., 2020).

Insomnia is characterized by symptoms indicating poor sleep quality, including difficulty falling asleep, unintended night awakenings, not feeling rested in the morning, daytime drowsiness, and impaired daytime functioning. Studies have shown that insomnia is highly prevalent among hemodialysis patients, with 40-83% experiencing sleep disturbances. These studies have found that sleep quality is low in hemodialysis patients, negatively impacting their quality of life, increasing cognitive impairment and inattentiveness, reducing work efficiency, and leading to higher mortality rates (Merlino et al., 2006; Al-Jahemodiyalizali et al., 2010; Hintistan et al., 2018; Rehman et al., 2020; Yang et al., 2021). In a study by Yıldırım et al. on insomnia, nearly all hemodialysis patients reported sleep problems both the night before (95.5%) and the night after (93.6%) dialysis treatment (Yıldırım et al., 2008). The frequent occurrence of sleep disorders and, consequently, insomnia during the hemodialysis process can be attributed to CKD-related biochemical and metabolic changes, lifestyle factors, other side effects of hemodialysis (such as fatigue, itching, and restless legs syndrome), as well as psychosocial issues like depression and anxiety (Özkan & Taylan, 2020).

Research on the effectiveness and safety of complementary and integrative therapies in treating HD complications is gaining increasing attention from researchers both nationally and internationally (Çevik & Taşçı, 2017; Eroğlu & Gök Metin, 2021; Suandika et al., 2023; Yeşil, 2023). The literature highlights that, in addition to pharmacological treatments, the use of non-pharmacological therapies in dialysis patients reduces fatigue, improves quality of life, enhances patient comfort, and is gaining increasing interest (Yeşil, 2023; Pompey et al., 2019; Sabouhi et al., 2013; Saeed et al., 2018; Yeşil Bayülgen & Gün, 2022). Among non-pharmacological treatment methods, acupressure, relaxation exercises, massage, reiki, and yoga can be independently performed by nurses, whereas aromatherapy, music therapy, and reflexology require physician supervision according to regulations (T.C. Traditional and Complementary Medicine Applications, 2014). Acupressure, a method from Traditional Chinese Medicine, is a technique based on the doctrine of meridians and acupuncture points. Acupressure is a gentle, safe, and non-invasive intervention with no risk of bleeding (Liu et al., 2023). The broad contact surface, easily controlled frequency and duration, and flexible pressure during massage enable both healthcare professionals and patient families to apply the method independently (İlter & Ovayolu, 2022; Eroğlu & Gök Metin, 2021). Consequently, acupressure is frequently used as an adjunct therapy to alleviate HD complications. Several studies have reported the effectiveness and safety of acupressure in treating HD complications (Marthoenis et al., 2021; Sabouhi et al., 2013; Saeed et al., 2018; Yeşil Bayülgen & Gün, 2022; Winzeler & Ambühl, 2020).

There are no randomized controlled studies investigating the effect of acupressure on sleep quality in HD patients. To establish the impact of acupressure on HD patients, high-quality, randomized controlled studies with sufficient sample sizes are needed. By implementing acupressure in this study, independent nursing interventions will be supported, increasing nurses' awareness and contributions to their practice. Additionally, if our research findings are adopted as institutional policy by hospital administrations, they will serve as a guide for nurses' care practices.

Research Objective This study aims to determine the effect of acupressure on sleep quality in hemodialysis patients.

Research Hypothesis H0: Acupressure has no effect on sleep quality in hemodialysis patients. H1: Acupressure has an effect on sleep quality in hemodialysis patients. Aim and Type of the Study This study is designed as a prospective, single-blind, randomized controlled trial to determine the effect of acupressure on sleep quality in hemodialysis (HD) patients. The study has been prepared based on the 25-item checklist and flowchart in the "Consolidated Standards of Reporting Trials (CONSORT-2017)." The Clinical Trials protocol registration will be completed via ClinicalTrials.gov.

Study Setting and Duration The study will be conducted at Adana City Training and Research Hospital Hemodialysis Unit between May 2025 and September 2025. In this dialysis unit, there are 110 patients receiving HD treatment three times a week on either Monday, Wednesday, and Friday or Tuesday, Thursday, and Saturday. The dialysis unit operates in three four-hour sessions daily, except on Sundays. The unit has a total of 40 dialysis machines. Patients diagnosed with Hepatitis B and Hepatitis C receive dialysis treatments in separate rooms with dedicated machines. The dialysis unit is ventilated through a central air conditioning system. The treatment areas provide appropriate conditions in terms of lighting, sound, privacy, and cleanliness, making them suitable for acupressure application. No complementary or integrative therapies aimed at reducing patient fatigue or improving quality of life and comfort are currently implemented in this unit.

Randomization A list of participants meeting the study criteria will be prepared by an independent researcher who is not involved in the study. After obtaining informed consent from patients willing to participate, their allocation to the intervention or control group will be determined randomly using the randomizer.org website. The 60 participants will be listed from 1 to 60, and the program will randomly assign them to one of two groups of 30 individuals each. The randomization process will be conducted by an independent researcher, ensuring that participants are randomly numbered by the system (randomizer.org).

Blinding Due to the nature of the study, the researcher will not be blinded, making this a single-blind, randomized controlled trial. After the study is completed, data will be entered into a computer by an independent researcher using "A" and "B" codes without specifying whether the data belongs to the intervention or control group. Data analysis and the preparation of the study report will be conducted by a statistician who is unaware of the group allocations, analyzing the data coded as "A" and "B." Data Collection Tools The study data will be collected using the "Patient Information Form" and the "Pittsburgh Sleep Quality Index (PSQI)." Patient Information Form: This form was created by the researcher based on a literature review to determine the socio-demographic characteristics of the participants. It consists of nine questions regarding age, gender, marital status, education level, income level, occupation, duration of HD treatment (in months/years), vascular access route, and the presence of any secondary disease.

Pittsburgh Sleep Quality Index (PSQI): Developed by Buysse et al. (1989), this self-report assessment tool provides information on sleep quality and the type and severity of sleep disturbances over the past month. The Turkish validity and reliability of the PSQI were established by Ağargün (1996). The PSQI consists of 19 self-reported questions and five additional questions answered by a bed partner or roommate, totaling 24 questions. It evaluates seven components: global sleep quality, subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each component is scored between 0 and 3, with the global PSQI score ranging from 0 to 21. Higher scores indicate poorer sleep quality and a higher level of sleep disturbance. A global PSQI score of 5 or above indicates clinically significant poor sleep quality (Buysse et al., 1989; Ağargün, 1996).

Implementation of Data Collection Tools The study consists of two groups: intervention and control. Patients meeting the study criteria will be informed about the study at the Adana City Training and Research Hospital Hemodialysis Unit. Those who agree to participate will sign informed consent forms, and the data collection forms will be administered. The intervention group will receive acupressure in addition to routine nursing care, while the control group will continue receiving routine nursing care without any additional intervention.

Application Bed and Support Pillows:

The application bed should neither be too hard nor too soft, and its dimensions should ensure the comfort of both the patient and the practitioner. A cylindrical pillow measuring 10-15 cm in diameter and 65-70 cm in length will be placed under the knees for support, along with an additional pillow for head support.

Application Position:

The patient will be positioned supine, with head and knee support provided by pillows, ensuring a comfortable and relaxed posture during the acupressure application.

Application Principles:

Acupressure will be applied by Specialist Nurse VDG, following the standards formulated by the World Health Organization. Hand hygiene will be maintained before and after each session. The acupressure points will be applied in the following order: Stomach 36 (ST 36), Gall Bladder 34 (GB 34), Spleen 6 (SP 6), and Kidney 1 (K 1). Care will be taken to ensure appropriate pressure intensity and duration, adjusting to individual sensitivity to prevent tissue damage. The pressure will be applied manually, using the thumb, index, and/or middle finger as appropriate for each anatomical location. The pressure will be applied at a frequency that is non-painful, non-disruptive, and has a calming effect.

Application Frequency, Timing, and Duration:

Based on previous studies (Liu et al., 2023; Suandike et al., 2023), acupressure will be applied three times a week for four weeks during the first two hours of HD sessions. The selected acupressure points include Stomach 36 (ST 36), Gall Bladder 34 (GB 34), Spleen 6 (SP 6), and Kidney 1 (K 1). Each session will target a total of eight points (four on each lower extremity). Before applying pressure, a preparatory warming rub will be performed for 10-15 seconds. Each point will receive approximately 90 seconds of pressure, totaling 12 minutes of application across all eight points. Including preparation, each session will last approximately 20 minutes.

Study Flow Process

Phase 1 (Preparation Phase):

An appropriate environment will be arranged in the Hemodialysis Units of Adana City Training and Research Hospital for patients in both the intervention and control groups.

Phase 2 (Implementation Phase):

This phase consists of four steps:

Eligible patients will be provided with brief information about the study, and their written informed consent will be obtained.

Patients meeting the inclusion and exclusion criteria will be selected, followed by the randomization process to form two groups. Participants will complete the "Informed Consent Form," "Patient Information Form," and "Pittsburgh Sleep Quality Index (PSQI)." Routine nursing care will be provided to both groups.

The intervention group will receive acupressure administered by Specialist Nurse Vecihe DÜZEL GÜNDÜZ, who has received training and certification in acupressure, for four weeks during the first two hours of HD, three times a week. The control group will receive only routine nursing care.

After four weeks, both groups will complete the "Pittsburgh Sleep Quality Index (PSQI)" again. To eliminate ethical concerns, acupressure will be offered to control group patients upon completion of the study.

Phase 3 (Reporting Phase):

Statistical analysis will be conducted on the collected data, and the study report will be prepared.

Ethical Considerations The study will be conducted in accordance with the Declaration of Helsinki. Ethical approval will be obtained from the Mersin University Clinical Research Ethics Committee, and written research permission will be obtained from the Adana Provincial Health Directorate. Written permission will be obtained from the developers of the scales used in the study. Participation will be voluntary, and confidentiality principles will be strictly followed. Patients will be informed that they can withdraw at any time, and all collected data will be securely stored by the researcher to ensure confidentiality.

Data Analysis The study data will be analyzed using appropriate statistical methods. Depending on the normality of data distribution, parametric or non-parametric tests will be applied for comparative data analysis. Descriptive statistics, including frequencies and percentages, will be provided. For normally distributed data, mean and standard deviation values will be presented, while for non-normally distributed data, minimum, maximum, median, and interquartile ranges (25th-75th percentiles) will be reported.

References Ağargün, M. Y., Kara, H., & Anlar, O. (1996). The validity and reliability of the Pittsburgh Sleep Quality Index. Turk Psikiyatri Derg, 7(2), 107-115.

Al-Jahemodiyalizali, H. H., Khogeer, H. A., Al-Qadhi, W. A., Baharoon, S., Tamim, H., Al-Hejaili, F. F., ... & Al-Sayyari, A. A. (2010). Insomnia in chronic renal patients on dialysis in Saudi Arabia. Journal of Circadian Rhythms, 8(1), 1-7.

Ammirati, A.L. (2020). Kronik böbrek hastalığı. Revista da Associação Médica Brasileira, 66, 3-9.

Buysse, D.J., Reynolds, C.F., Monk, T.H., Berman, S.R., Kupfer, D.J., 1989. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 28(2):193-213.

Çevik, B., Taşcı, S. (2017). Akupres uygulamasının ağrı yönetimine etkisi. Sağlık Bilimleri Dergisi, 26(3), 257-261.

Eminsoy, İ. O. (2018). Renal Replasman Tedavisi Alan Yetişkin Hastaların Tıbbi Beslenme Tedavisi: Bir Olgu Sunumu. Beslenme ve Diyet Dergisi, 46, 94-99.

Eroğlu, H., Gök Metin, Z. (2021). Hemodiyaliz hastalarında semptom yönetiminde tamamlayıcı ve integratif yaklaşımlar: Sistematik bir derleme. Hacettepe Üniversitesi Hemşirelik Fakültesi Dergisi, 8(3), 252 - 268.

Hintistan, S., & Deniz, A. (2018). Hemodiyaliz tedavisi alan hastalarda semptom değerlendirmesi. Bezmialem Science, 6, 112-8.

İlter, S.M., Ovayolu, Ö. (2022). Hemodiyaliz hastalarının yorgunluk yönetiminde kanıta dayalı integratif yaklaşımlar. Hacettepe Üniversitesi Hemşirelik Fakültesi Dergisi, 9(1), 82-88., Kalantar-Zadeh, K., Jafar, T. H., Nitsch, D., Neuen, B. L., & Perkovic, V. (2021). Chronic kidney disease. The Lancet, 398(10302), 786-802.

Liu, C., Yang, J., Li, H., He, P., Deng, Y., Dong, A., Ma, Y., Zhang, S., Chen, S., Zhang, M. (2023). Acupressure for sleep disorders, fatigue, depression and pruritus in hemodialysis patients: A systematic review and meta-analysis. Research Square. 1,1-14.

Marthoenis, M., Syukri, M., Abdullah, A., Tandi, T. M. R., Putra, N., Laura, H., Setiawan, A., Sofyan, H., Schouler-Ocak, M. (2021). Quality of life, depression, and anxiety of patients undergoing hemodialysis: Significant role of acceptance of the illness. International Journal of Psychiatry in Medicine, 56(1), 40-50.

Merlino, G., Piani, A., Dolso, P., Adorati, M., Cancelli, I., Valente, M., & Gigli, G. L. (2006). Sleep disorders in patients with end-stage renal disease undergoing dialysis therapy. Nephrology Dialysis Transplantation, 21(1), 184-190.

Özkan, İ., & Taylan, S. Hemodiyaliz Hastalarında Kaşıntının Varlığı ile Uyku ve Anksiyete Arasındaki İlişkinin İncelenmesi. Nefroloji Hemşireliği Dergisi, 15(2), 66- 78.

Pompey, C. S., Ridwan, M. N., Zahra, A. N., Yona, S. (2019). Illness acceptance and quality of life among end state renal disease patients undergoing hemodialysis. Enfermeria Clinica, 29, 128- 133.

Rehman, O. F., Rauf, U., Rauf, M., Aziz, S., Faraz, A., & Jameel, F. A. (2020). Association of Insomnia in Patients with Chronic Kidney Disease on Maintenance Hemodialysis. Cureus, 12(8).

Sabouhi, F., Kalani, L., Valiani, M., Mortazavi, M., Bemanian, M. (2013). Effect of acupressure on fatigue in patients on hemodialysis. Iranian Journal of Nursing and Midwifery Research, 18(6), 429-434.

Saeed, S., Islahudin, F.H., Bakry, M.M., Redzuan, A.M. (2018). The practice of complementary and alternative medicine among chronic kidney disease patients. Journal of Advanced Pharmacy Education Research, 8 (3), 30-36.

Suandika, M., Chen, S. Y., Fang, J. T., Yang, S. H., Tsai, Y. F., Weng, L. C., Tsay, P. K., Tang, W. R. (2023). Effect of acupressure on fatigue in hemodialysis patients: A single-blinded randomized controlled trial. Journal of İntegrative and Complementary Medicine, 29(2), 111-118.

T.C. Geleneksel ve Tamamlayıcı Tıp Uygulamaları (2014). Geleneksel ve Tamamlayıcı Tıp Uygulamaları Yönetmeliği. T.C. Resmi Gazete; 2014 Ekim 27. No. 29158. 10 Eylül 2023 tarihinde URL:http://www.resmigazete.gov.tr/eskiler/2014/10/20141027- 3.adresinden erişildi Tolasa, A. G., & Akyol, A. Diyaliz Hastalarında Aromaterapi Kullanımı. Nefroloji Hemşireliği Dergisi, 12(2), 84-90.

Tuna, D., Ovayolu, N., & Duygu, K. (2018). Hemodiyaliz hastalarında sık karşılaşılan problemler ve çözüm önerileri. Nefroloji Hemşireliği Dergisi, 13(1), 17-25.

Turgay, G., Eler, Ç. Ö., Ökdem, Ş., &Kaya, S., (2020). Hemodiyaliz hastalarında progresif gevşeme egzersizinin konfor düzeyine etkisi. Nefroloji Hemşireliği Dergisi, 15(1), 16-22.

Webster, A. C., Nagler, E. V., Morton, R. L., & Masson, P. (2017). Chronic kidney disease. The lancet, 389(10075), 1238-1252. https://Doi.org/10.1016/S0140- 6736(16)32064-5 Winzeler, R., Ambühl, P. M. (2020). P1467 Demography of the dialysis population in Swıtzerland in 2018. Nephrology Dialysis Transplantation, 35(3), 142.

Yang, X. X., Hao, L. Y., Chen, Y. Y., & Meng, F. J. (2021). Effects of progressive muscle relaxation therapy on Maintenance Hemodialysis patients: a systematic review and meta-analysis. TMR Integrative Medicine, 5, e21003.

Yeşil Bayülgen M. (2023). Examination of graduate nursing thesis regarding the symptom of fatigue in dialysis patients. Black Sea Journal of Health Science, 6(4),564-570.

Yeşil Bayülgen M., Gün, M. 2022. Effect of complementary and ıntegrative treatments on fatigue symptoms in hemodialysis patients. Holistic Nursing Practice, 36(1),17-27.

Yıldırım, Y., Akyol, A. D., & Fadıloğlu, Ç. (2008). Hemodiyaliz Tedavisi Gören Son Dönem Böbrek Yetmezliği Hastalarında Uyku Sorunları. Nefroloji Hemşireliği Dergisi, 5(1-2), 31-37.

Yılmaz, F. T., Sert, H. Kumsar, A. K., Aygin, D., Sipahi, S., & Genç, A. B. (2020). Hemodiyaliz Tedavisi Alan Hastaların Umut Düzeyleri, Semptom Kontrolü ve Tedaviye Uyumlarının Değerlendirilmesi. Acıbadem Üniversitesi Sağlık Bilimleri Dergisi, (1), 35-43.

ELIGIBILITY:
Inclusion Criteria:

* Informed Voluntary Consent Form/Written Consent Form signed by the patient
* Able to read, write, speak and understand Turkish
* Over 18 years of age
* Receiving HD treatment for at least 6 months
* Receiving HD treatment 3 times a week
* Conscious, fully oriented and cooperative, and open to communication
* No vision, hearing and perception problems
* General condition good and comfortable (vital signs within normal limits)

Exclusion Criteria:

* Patients who do not sign the Informed Consent Form/Written Consent Form
* Those who cannot read, write or understand Turkish
* Those who are under 18 years of age
* Those who have received HD treatment for less than 6 months
* Those who receive HD treatment twice a week
* Those who are unconscious, have incomplete orientation and cooperation and are closed to communication
* Those who have vision, hearing and perception problems
* Those whose general condition is not good
* Those who have a wound or amputation in the lower extremity, rheumatoid arthritis or limb fracture
* Those who have any psychiatric disease
* Those who have Hepatitis B and Hepatitis C
* Those who use any of the complementary and integrated methods

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality: This measure will assess the quality of sleep during the intervention period. | It will be measured twice: the first test at the first meeting with the patient and the final test four weeks later.
  The PSQI scale will be recorded to assess the individual's sleep quality, quantity, presence and severity of sleep disturbance.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) in this study